CLINICAL TRIAL: NCT06819904
Title: Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE) for mTBI: A Targeted Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE) RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Research Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24040027; HT94252320064 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-05-06; First posted 2025-02-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Mild; Mild Traumatic Brain Injury (mTBI); Vestibular; Psychological Health
Keywords: concussion; mTBI; vestibular; psychological health
MeSH Terms: conditions — Brain Concussion; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The current study will employ a single blinded, two-group repeated measures (baseline, 4-week, 3-month, 6-month) design with permuted block random assignment to ACTIVE and Vestib Control groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE) (Experimental): The ACTIVE intervention group will receive Acceptance and Commitment Therapy (ACT) + targeted vestibular rehabilitation exercises and behavioral management during four weekly in person sessions along with daily at-home activities during the 4 week treatment period. The four ACTIVE sessions will last 90 minutes and will be divided between the vestibular rehabilitation portion (30 minutes) and the ACT portion (60 minutes). ACT component and therapy sessions will include: 1) values clarification and goal setting; 2) skills training in psychological flexibility including emotional acceptance, cognitive defusion, and present moment awareness; and 3) practice engaging these skills to overcome mental obstacles to values-driven goal attainment.
  Interventions: Behavioral: Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE)
- Usual Care Vestibular Rehabilitation (VESTIB CONTROL) (Active Comparator): The VESTIB CONTROL group will receive standard of care evaluations and treatments involving a holistic multidisciplinary approach, which includes vestibular rehabilitation, but will exclude any ACT components. Because usual standard of care is individualized to the patient's unique functional deficits, treatments combined with vestibular rehabilitation may focus on any one or more of the following: neuro-optometry, neuropsychology, physical and occupational therapy, or speech and language pathology, or general mental health interventions such as instruction regarding stress reduction. Participants will attend 4 weekly in-person visits for vestibular rehab, as well as any other interventions provided to them by their treating clinician.
  Interventions: Behavioral: Usual Care Vestibular Rehabilitation

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE) — Participants will receive the ACT treatment. It is comprised of three processes: Open Up, Be Present, and Do What Matters. Each of these is further sub-divided, for a total of six core processes. These processes include, but are not limited to, present moment awareness, de-fusion, and committed action. This group will also receive targeted vestibular therapy and standardized behavioral management strategies (physical activity, sleep, hydration, and nutrition prescription). Participants will also receive usual care at the discretion of each site's treating providers. They will also receive vestibular therapy that may include one or more exercises in the following groups: 1) gaze stability, 2) visual-vestibular habituation, and 3) balance/gait.
  Arms: Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE)
Behavioral: Usual Care Vestibular Rehabilitation — Participants will receive usual care at the discretion of each site's treating providers, excluding any components associated with ACT. They will also receive vestibular therapy that may include one or more exercises in the following groups: 1) gaze stability, 2) visual-vestibular habituation, and 3) balance/gait.
  Arms: Usual Care Vestibular Rehabilitation (VESTIB CONTROL)

SUMMARY:
The primary objective of this multi-site randomized clinical trial (RCT) is to compare Acceptance and Commitment Therapy Integrated Vestibular Rehabilitation (ACTIVE) with usual care vestibular rehabilitation (VESTIB CONTROL) in 250 individuals with mTBI-related vestibular symptoms attributable to mild traumatic brain injury (mTBI) treated at one of two sites (1) the University of Pittsburgh Medical Center, or (2) the Intrepid Spirit Center, Carl R. Darnall Army Medical Center, Fort Hood, Texas. Both interventions will be delivered weekly over 4 weeks. Assessments will be administered prior to the start of treatment (Baseline) and at 4-weeks, 3- and 6-months following the completion of treatment.

DETAILED DESCRIPTION:
Nearly 378,000 mTBIs have occurred among U.S. military service members (SM) since 2000. These injuries result in myriad symptoms (e.g., dizziness, headache, fogginess) and impairments (e.g., cognitive, ocular, vestibular) that typically resolve within a month. However, many SMs experience symptoms and impairment lasting months or longer, resulting in limited operational readiness and duty restrictions. As such, one of the challenges related to mTBI and psychological health issues in military SMs is identifying and implementing timely and effective treatments that address these symptoms in an integrated manner and mitigate downstream problems.

Interventions are needed to target comorbid mTBI and psychological health symptoms. Previous research suggests that targeted vestibular rehabilitation combined with behavioral management (physical activity, sleep, nutrition, hydration) is effective in improving vestibular symptoms and associated functional impairment and reducing recovery time following mTBI. Acceptance and Commitment Therapy (ACT) is a trans-diagnostic cognitive-behavioral therapy based on incorporation of mindfulness and acceptance-based work into traditional behavior therapy. ACT is designed to improve psychological health, functioning, and well-being by improving psychological flexibility or the ability to remain present in the moment despite emotional distress.

There is separate evidence for the effectiveness of targeted vestibular rehabilitation combined with behavioral management interventions, and ACT in regard to enhancing recovery from mTBI and PH, respectively. However, researchers have yet to synergize these approaches to evaluate their effectiveness in military SMs following mTBI involving vestibular and psychological health domains. Our overarching hypothesis is that a combined, brief (<4 weeks) intervention involving both ACT and integrated vestibular rehabilitation (ACTIVE) will reduce symptoms, impairment, and functional limitations, and accelerate return to activity among military SMs and civilians following mTBI with vestibular symptoms/impairment compared to usual care vestibular rehabilitation (VESTIB CONTROL). The investigators believe that the potential synergy of these combined interventions could provide a more efficient and effective treatment strategy that could mitigate downstream psychological health morbidity in the estimated 60-65% of SMs with vestibular symptoms and impairment following mTBI.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years of age
* Normal/corrected vision
* Diagnosed with mTBI per military clinical practice guidelines (CPGs) that occurred over 8 days prior to consent as determined by a multi-domain assessment performed by a licensed healthcare professional.
* Reported or observed signs of mTBI including loss of consciousness, amnesia, disorientation/confusion, dizziness, imbalance, memory problems, vomiting at the time of injury as determined by self-report.
* Positive for mTBI-related vestibular symptoms and/or impairments per a concussion common data elements (CDE) assessment. Participants must demonstrate a positive finding in at least one of the following tests: DVAT (>2 lines lost), DNRS (>2/10 score), VVAS (>0 on 2 or more items), VOMS (>2 score on VOR or VMS), mBESS (> 9 total errors), and CP-Screen (avg vestibular factor score >/= 2 or single item = 3 severity)

Exclusion Criteria:

* History of vestibular disorder (e.g., benign paroxysmal positional vertigo, unilateral or bilateral vestibular hypofunction) as determined by patient self-report and/or by Physical Therapist exam.
* Exercise-induced dizziness as determined by the Physical Therapist exam.
* History of neurological disorder (e.g., epilepsy, multiple sclerosis) as determined by self-report.
* Cervical spine injury or dysfunction (i.e., limited range of motion; ROM) as determined by self-report.
* Previous moderate to severe TBI as determined by self-report.
* < 8 days following current mTBI as determined by self-report.
* Currently pregnant as determined by self-report.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline, 4-week, 3-month, 6-month study visits
  The DHI is a 25-item self-report measure that examines dizziness-related handicap. Each item is categorized into one of three domains: functional, emotional, or physical. The DHI was developed with the help of patients who complained of dizziness and uses a three-item response scale (Yes, Sometimes, No) scored as 4/2/0, respectively. Score range: 0-100, with higher scores indicating worse dizziness.
Generalized Anxiety Disorder (GAD-7) | Baseline, 4-week, 3-month, 6-month study visits
  The GAD-7 is a seven item self-reported questionnaire that measures severity of symptoms regarding anxiety. Responses are 0 = not at all, 1 = several days, 2= more than half the days, and 3 = nearly every day. Higher scores are indicative of higher anxiety (0-4 = minimal anxiety, 5-9= mild anxiety, 10-14 =moderate anxiety, 15-21 = severe anxiety.

SECONDARY OUTCOMES:
Ohio State University TBI Identification short form (OSU TBI-ID) | Baseline
  The OSU TBI-ID is a standardized form that collects lifetime instances of brain injuries via a 3-5 minute structured interview. For each past reported instance of a brain injury, the form collects the mechanism of injury, the occurrence of loss of consciousness (yes/no), duration of loss of consciousness (< 30 mins, 30min-24hr, >30 min), became dazed or experienced a memory gap, and age at injury.
Dynamic Visual Acuity Test (DVAT) | Baseline
  The DVAT is a functional evaluation tool for the impairment and compensation of the vestibular system, which could reflect the Vestibulo-ocular reflex (VOR) function. Static (i.e., no head movement) visual acuity is measured first by having the individual sit 20 feet from standard optometric Snellen Chart and read the lowest line recognizable. The physical therapist will then gently grasp the individual's head and oscillate them back and forth (20-30 degrees from midline at 2Hz). The individual will then read the lowest line possible. A loss of 3 lines or more of visual acuity relative to their static visual acuity is regarded as clinically significant and suggestive of possible vestibular dysfunction.
Dizziness Numerical Rating Scale (DNRS) | Baseline
  The Defense and Veterans Pain Rating Scale (DVPRS) was created to standardize pain reporting and measurement across the military. It will be adapted for use specifically for dizziness. Changes to the verbal anchors include: 0 = "no dizziness", 1 = "hardly notice dizziness", 2 = "Notice dizziness, does not interfere with activities", 9 = "can't bear the dizziness, unable to do anything", 10 = "As bad as it could be, nothing else matters". Participants will be asked for their current dizziness during the past week, with higher scores indicating worse dizziness. The DNRS takes 1 minute to administer, and used in the screening process.
Visual Vertigo Analog Scale (VVAS) | Baseline
  The VVAS assesses how much dizziness 0 (none) to 10 (severe), on a visual analog scale, an individual reports for 9 different activities, such as walking through a supermarket aisle, being in a room with fluorescent lights, doing down and escalator, walking over a patterned floor, etc. A positive result (indicating more dizziness symptoms) occurs when an individual rates at least two of the nine items of the VVAS above zero (VVAS positive). The VVAS takes 5 minutes to administer, and used in the screening process.
Concussion Clinical Profiles Screening (CP-Screen) | Baseline
  The CP Screen is a 29 item self-report, clinical profiles based symptom inventory that measures five concussion clinical profiles: 1) anxiety/mood, 2)cognitive/fatigue, 3) migraine, 4) ocular, 5) vestibular; and two modifying factors sleep and cervical. Participants indicate on a scale of 0 (none) to 3 (severe) the level of symptom severity for each item. The CP screen yields an average factor and modifier scores, with higher scores indicative of worse symptom severity, score range is 0-87.
Vestibular/Ocular Motor Screening (VOMS) - Change from Baseline in Symptom Reporting at 4-weeks | Baseline, 4-week
  The VOMS assesses impairment via patient-reported symptom provocation following each of the following items: 1) smooth pursuits; 2) horizontal and vertical saccades; 3) convergence; 4) horizontal and vertical ocular reflex (VOR); and 5) visual motion sensitivity (VMS).
  Patients rate their symptom severity in headache, dizziness, nausea, and fogginess compared to their immediate pre-assessment state on a scale of 0 (none) to 10 (severe) to determine if any VOMS item provokes the symptoms. Scores on any symptom of 2 or greater reflects a positive screening cut-off for vestibular or oculomotor impairment. Total symptom scores are recorded for each symptom.
  Scores will be compared between Baseline and 4-week visits
Vestibular/Ocular Motor Screening (VOMS) - Change from Baseline in Convergence Measurement at 4-Weeks | Baseline, 4-week
  See Outcome 8 for description of VOMS test.
  Convergence is also assessed in the VOMS using objective measurement of the near point of convergence (NPC). It is averaged across 3 trials, and recorded in centimeters (cm). NPC values >5 cm reflect a positive clinical screening.
  Scores will be compared between Baseline and 4-week visits
Modified Balance Error Scoring System (mBESS) - Change from Baseline in Total Errors at 4-weeks | Baseline, 4-week
  The mBESS measures postural stability and consists of three stances including feet side by side, a tandem stance, and a single-leg stance on the non-dominant leg. The three stances are performed for 20 seconds each on a firm surface. All stances are completed with eyes closed and with hands on the iliac crests. Errors include lifting hands off the iliac crests, opening the eyes, stepping, stumbling, falling, moving the hips more than 30 degrees of flexion or abduction, lifting the forefoot or heel, or remaining out of the testing position for more than 5 seconds. Each error equals 1 point, with higher scores indicating worse performance. For the current study, the modified BESS (mBESS) on the firm surface only will be used. Clinical cut-offs for mBESS suggest a total error of 9 or greater indicate clinical impairment in balance. The mBESS takes approximately 5-6 minutes to administer. mBESS scores will be analyzed at each timepoint and over time.
Neurobehavioral Symptom Inventory (NSI) | Baseline, 4-week, 3-month, 6-month study visits
  The NSI is a 22-item symptoms scale in which participants rate the severity of symptoms on a 5-point scale (0=none, 1= mild, 2=moderate, 3=severe, 4=very severe) Scores range from 0 to 60. The NSI takes approximately 5-10 minutes to administer. NSI total score changes will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
Patient Health Questionnaire 9 (PHQ-9) | Baseline, 4-week, 3-month, 6-month study visits
  The PHQ-9 is a 9 item questionnaire that assesses the presence and severity of depression. Total score ranges from 1-27, with higher scores indicating higher level of depression. Scale is 0-4 (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day). PHQ-9 total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
DSM-Cross Cutting Symptom Measure - Adult (DSM-CCSM-A) | Baseline, 4-week, 3-month, 6-month study visits
  The DSM-CCSM-A is a 23-item self-report measure designed to evaluate overall and co-occurring psychological health symptoms including depression, anger, mania, anxiety, somatic symptoms, sleep disturbance, psychosis, obsessive thoughts/behaviors, substance use, personality function, dissociation, cognition, and suicide. The DSM-CCSM-A is commonly used to track therapeutic response to interventions. All items except for the three suicide-related items are rated 0-none to 4-severe/almost daily. Items scored at 2 or greater indicate important levels of symptoms that require further assessment. Scores range from 0-88. Scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
PTSD Checklist (PCL-5) | Baseline, 4-week, 3-month, 6-month study visits
  The PCL-5 is a 20-item self-report questionnaire corresponding to the DSM-5 symptom criteria for PTSD. The wording of PCL-5 items reflects both changes to existing symptoms and the addition of new symptoms. The items are rated on a 5-point Likert scale, 0-4 for each symptom, and summed for a total severity score ranging from 0-80. Total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
World Health Organization Disability Assessment Schedule 2 (WHODAS 2.0) | Baseline, 4-week, 3-month, 6-month study visits
  The WHODAS 2.0 Measures average functioning in everyday situations over the last 30 days, and surveys six domains of functioning (cognition, mobility, self-care, getting along with others, life activities and participation. The modified version will be used in this study. It contains 12 items rated on a 5-point scale 0-4, with summary score of 0-100 (where 0 = no disability; 100 = full disability). Total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
Acceptance and Action Questionnaire - Version 2 (AAQ-II) | Baseline, 4-week, 3-month, 6-month study visits
  The AAQ-II is a 7-item self-report questionnaire with items rated on a 7-point Likert scale 1-7 (1=Never true to 7=Always true). It is used to measure an individual's behaviors regarding their ability to process feelings, emotions, and worries. It is often used to measure progress in Acceptance and Commitment Therapy. Higher total scores indicate higher psychological inflexibility, experiential avoidance, and more potential psychological distress. Total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
Work and Social Adjustment Scale (WSAS) | Baseline, 4-week, 3-month, 6-month study visits
  The WSAS assesses the impact of a person's mental health difficulties on their ability to function in terms of work, home management, social leisure, private leisure and personal or family relationships. It is a 5-item self-report questionnaire on a 9-point Likert scale 0-8 (0=Not at all; 8=Very Severely). Higher scores indicate greater difficulty. Total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
Patient Global Impression of Change (PGIC) | 4-week, 3-month, 6-month study visits
  The PGIC was developed for self-reported assessment of change resulting from post-concussion care at military treatment facilities. The prompt is: ""Since beginning treatment at this facility, how would you describe the change (if any) in ACTIVITY LIMITATIONS, SYMPTOMS, EMOTIONS and OVERALL QUALITY OF LIFE related to your post-concussive condition?"" The participant responds on a scale ranging from 0 (No change or condition has gotten worse), to 7 (A great deal better and a considerable improvement that has made all the difference). Lower scores indicate worse recovery. Total scores will be analyzed between Baseline to 4-weeks to 3-months and to 6-months.
Return to Duty (RTD)/Return to Activity (RTA) Status | Baseline, 4-week, 3-month, 6-month study visits
  For civilians, return to activity (RTA) will be medical clearance to resume full activities without limitations based on symptom and impairment free at rest, and symptom free following standardized exertion protocols per recent consensus. Return to duty (RTD) will be determined based on: Not returned to duty/Returned to duty with restrictions/Returned to duty without restrictions.
I-Portal Portable Assessment System (I-PAS) - Eye Movements | Baseline, 4-week
  Description of test: The I-PAS is a portable, 3-D virtual reality (VR)-based, video-oculographic test device to evaluate vestibulo-ocular function. The goggles are placed on the head of participants who are then asked to follow the instructions on the VR display. A series of vestibulo-ocular tests are performed, and data is recorded via laptop interface. Participants will perform the following static and dynamic vestibular tests: spontaneous nystagmus, gaze nystagmus, positional, sinusoidal harmonic acceleration (SHA), SHA with visual enhancement and suppression; head impulse tests; as well as vestibulo-ocular and oculomotor tests including: smooth pursuits, vergence pursuit, vergence steps, predicted saccades, anti-saccades, visual vertical and horizontal, visual reaction time, and dual eye movement/motor tasks.
  The eye movements of each tested are recorded, and the changes in movement will be assessed from baseline to 4-week.
I-Portal Portable Assessment System (I-PAS) - Symptoms | Baseline, 4-week
  Please see description of I-PAS test in Outcome 19.
  Symptom severity will be rated 0 (none) to 10 (severe) for headache, nausea, dizziness, and fogginess before and after the I-PAS testing procedures. The totals will be compared from the beginning of the test to after, as well as between visits.
Fitbit Activity | Daily, starting at Baseline and ending at 4-week
  At Baseline, the study team will provide all participants with a Fitbit Inspire 3 (or similar device depending on market availability) physical activity tracker to wear and sync with participant's cell phones for the duration of the 4-week intervention period. The activity monitoring will provide confirmatory evidence of compliance via real-time monitoring of physical activity and sleep behaviors.
  The study team will download the Fitbit data collected, such as (but not limited to) step counts, heart rate, sleep, and daily activity across each day of the 4-week intervention period from Fitabase.
Fitbit Activity - Step Counts | Daily, starting at Baseline and ending at 4-week
  See Outcome 22 for description of Fitbit
  Daily step counts will be recorded.
Fitbit Activity - Heart Rate | Daily, starting at Baseline and ending at 4-week
  See Outcome 22 for description of Fitbit
  Daily heart rate (HR) measured as beats per minute will be recorded. This will include daily average, hour average, and minute average.
Fitbit Activity - Sleep | Daily, starting at Baseline and ending at 4-week
  See Outcome 22 for description of Fitbit
  Daily sleep information will be recorded. For each day/night of sleep, the following will be recorded: 1)minutes asleep, 2) minutes after wakeup, 3) minutes to fall asleep, 4) minutes of time in bed.
Fitbit Activity - Daily Activity | Daily, starting at Baseline and ending at 4-week
  See Outcome 22 for description of Fitbit
  Daily activity information will be recorded. For each day of activity, the following is recorded: 1)distance walked (miles), 2) time of activity (minutes), 3) calories burned

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Concussion Research Laboratory, Pittsburgh, Pennsylvania
  - Intrepid Spirit Center, Carl R. Darnall Army Medical Center, Fort Hood, Texas

IPD SHARING:
Plan to Share IPD: Yes
Per DoD grant requirement, de-identified data will be shared with the Federal Interagency Traumatic Brian Injury Research (FITBIR) informatics system and Congressionally Directed Medical Research Programs (CDMRP). This data includes non-identifiable demographic data, medical history, medications, and both primary and secondary outcomes (except I-PAS and Fitbit data).
Time Frame: De-identified data will be shared with FITBIR on an annual basis as required by the funder (DoD). Data will be entered until the study has completed. All data will be available on the FITBIR website indefinitely.
Access Criteria: Formal requests must be submitted and approved to FITBIR to access this study's de-identified data.
URL: https://fitbir.nih.gov